CLINICAL TRIAL: NCT02606708
Title: Accelerated Intensity Modulated Radiation Therapy (AIMRT) to the Breast After Segmental Mastectomy: a Pilot Study
Brief Title: Accelerated Intensity Modulated Radiation Therapy (AIMRT) to the Breast After Segmental Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11105
Record Dates: First submitted 2015-09-30; First posted 2015-11-17 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated intensity modulated radiation therapy (AIMRT) (Experimental): All patients shall receive a total of 40.5 Gy to the entire breast in 2.7 Gy/fraction x 15 fractions, Monday to Friday for 3 weeks delivered prone in uniform daily doses through IMRT tangent fields. A concurrent boost to the original tumor bed of 0.50 Gy will be delivered.
  Interventions: Radiation: Accelerated intensity modulated radiation therapy (AIMRT)

INTERVENTIONS:
Radiation: Accelerated intensity modulated radiation therapy (AIMRT)

SUMMARY:
The primary purpose of this study is to determine the feasibility and tolerability of a regimen of accelerated (hypofractionated) Intensity Modulated Radiation Therapy (AIMRT) to the whole breast as part of breast preservation. In addition, the investigators want to prospectively collect blood specimens to: assess TGF-β polymorphisms to identify potential carriers at higher risk for post-treatment fibrosis; generate a blood specimen repository for future studies of other relevant polymorphisms. The study investigators also want to prospectively follow each treated woman yearly to assess long-term radiation sequelae of the current regimen by using the LENT/SOMA scores.

DETAILED DESCRIPTION:
Despite level I evidence of comparable efficacy to that of mastectomy, breast conserving therapy (BCT) remains underutilized in the United States. In 1990, the National Institutes of Health (NIH) Consensus Development Conference concluded that BCT was the appropriate method of treatment for the majority of women with early stage I and II breast cancer. However, this subsequently only translated in a moderate increase in the utilization of BCT, shifting from 34% to 60% for stage I breast cancer and from 19% to 39% for stage II breast cancer.

There appear to be multiple causes for underutilization. The demands of the standard radiation schedule probably play the main role. Generally, post-lumpectomy radiation therapy consists of 4 to 5 weeks of whole breast radiation of a total dose 45 to 50 Gy in 23-25 fractions, usually followed by a boost of 10 to 16 Gy in 5-8 fractions to the tumor bed area. The total length of treatment is 5-7 weeks, commonly six weeks. Practically, women who choose BCT automatically commit to a regimen of approximately six weeks of daily radiation visits (Monday to Friday) to complete the local management of their breast cancer. For many women, concerns about this commitment are likely to influence the choice for mastectomy instead of breast preservation since only 40-60% of women who meet criteria for BCT actually undergo the procedure. In addition to possible biases of the primary health care provider affecting these choices, it is known that distance from RT treatment facilities also plays an important role in women's choice for mastectomy instead of BCT. Unfortunately, 15-30% of patients who have actually selected BCT, in particularly older patients and those with 2 or more co-morbid conditions, do not receive postoperative RT. These facts warrant a critical assessment of standard radiation therapy in this clinical setting.

The actual standard approach to post-segmental mastectomy adjuvant radiation at our institution consists of surgical excision followed by 6 weeks of breast irradiation for a total of 30 fractions of 2 Gy each, 23 (46 Gy) to the whole breast while 7 to the original tumor bed (14 Gy). Instead, the women in this study will only receive 15 larger radiation fractions (2.7 Gy) to the entire breast with a concomitant boost to the tumor bed (2.7 Gy + .5 Gy, total 3.2 Gy per fraction). All women will be treated prone to best apply IMRT techniques while avoiding the rest of the body.

Treatment with fewer fractions over a shorter duration of time offers several advantages, provided it is as effective as the conventional treatment regimens and without added morbidity. The potential advantages include: 1) less time away from homes, families and jobs; 2) less cost associated with travel and time away from work; 3) ease the demand on radiation treatment resources and produce savings to the health-care system. Moreover, treatment prone assures that only minimal dose of radiation is delivered to the lung, heart and to the controlateral breast.

Patients will have completed all breast surgical procedures prior to accrual into this protocol in order to establish eligibility criteria. All patients will then be treated prone with 2.7 Gy/fraction delivered in 15 fractions over a 3-week period for a total dose of 40.5 Gy.

All patients will be followed 1, 3, 6, 12 months after treatment course, then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pre- or post-menopausal women with Stage I and II breast cancer
* Biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm
* Status post segmental mastectomy. and after sentinel node biopsy and/or axillary node dissection
* At least 2 weeks from last chemotherapy
* Tumors < 5 mm do not require nodal assessment

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast.
* More than 3 involved nodes identified at axillary staging, requiring adjuvant axillary radiation.
* Active connective tissue disorders, such as lupus or scleroderma.
* Prior or concurrent malignancy other than basal or squamous cell skin cancer or carcinoma in-situ of the cervix, unless disease-free > 5 years.
* Pregnant or lactating women.

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2005-02-20 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Accelerated Intensity Modulated Radiation Therapy (AIMRT): All patients shall receive a total of 40.5 Gy to the entire breast in 2.7 Gy/fraction x 15 fractions, Monday to Friday for 3 weeks delivered prone in uniform daily doses through IMRT tangent fields. A concurrent boost to the original tumor bed of 0.50 Gy will be delivered.
  Accelerated intensity modulated radiation therapy (AIMRT)
Period: Overall Study
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Started | 314
Completed | 314
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 188
  >=65 years | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 220
  Black | 60
  Asian | 22
  Hispanic | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 314

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Recurrence in Breast
Description: Defined by the discovery of invasive disease or DCIS in the same region of the breast after segmental mastectomy and radiation, by clinical or radiographic means.
Time Frame: 5 years
Population: Risk rate at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants | 6

2. Primary Outcome: Number of Participants With Regional Recurrence
Description: Defined by the discovery of invasive disease or DCIS regional recurrence in the lymph node after segmental mastectomy and radiation, by clinical or radiographic means.
Time Frame: 5 years
Population: Risk rate at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants | 4

3. Primary Outcome: Number of Participants With Contralateral Breast Cancer
Description: Defined by the discovery of contra-lateral breast cancer after segmental mastectomy and radiation, by clinical or radio-graphic means.
Time Frame: 5 years
Population: Risk rate at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants | 2

4. Primary Outcome: Number of Participants With Distant Metastases
Description: number of participants found to have distant metastases after segmental mastectomy and radiation, by clinical or radiographic means
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants | 8

5. Primary Outcome: Number of Participants With an Outcome of Death
Description: Overall 5-Year cumulative rate of death based on Kaplan-Meier Analysis
Time Frame: 5 years
Population: Risk rate at 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants | 17

6. Secondary Outcome: Maximum Grade Late Radiation Toxicity
Description: Measure of treatment related late toxicities at or more than 6 months after completion of radiation therapy.
Time Frame: 5 years
Population: Overall, 314 participants were analyzed for each of the below listed toxicities, by grade. The numbers are broken down to toxicity and grade for each row. In total these numbers add to 314
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants
  Pigmentation Change: number analyzed (Participants) | 64
  Pigmentation Change: Grade 1 | 62
  Pigmentation Change: Grade 2 | 2
  Pigmentation Change: Grade 3 | 0
  Breast Fibrosis: number analyzed (Participants) | 73
  Breast Fibrosis: Grade 1 | 59
  Breast Fibrosis: Grade 2 | 13
  Breast Fibrosis: Grade 3 | 1
  Breast Retraction: number analyzed (Participants) | 65
  Breast Retraction: Grade 1 | 46
  Breast Retraction: Grade 2 | 17
  Breast Retraction: Grade 3 | 2
  Breast Telangiectasia: number analyzed (Participants) | 70
  Breast Telangiectasia: Grade 1 | 47
  Breast Telangiectasia: Grade 2 | 19
  Breast Telangiectasia: Grade 3 | 4
  Breast Edema: number analyzed (Participants) | 11
  Breast Edema: Grade 1 | 10
  Breast Edema: Grade 2 | 0
  Breast Edema: Grade 3 | 1
  Breast Pain: number analyzed (Participants) | 29
  Breast Pain: Grade 1 | 28
  Breast Pain: Grade 2 | 1
  Breast Pain: Grade 3 | 0
  Arm Lymphadema: number analyzed (Participants) | 2
  Arm Lymphadema: Grade 1 | 1
  Arm Lymphadema: Grade 2 | 0
  Arm Lymphadema: Grade 3 | 1

7. Secondary Outcome: Patient Self-assessment of the Cosmetic Results
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
Participants
  Excellent/Good | 251
  Fair | 56
  Poor | 7

8. Secondary Outcome: Survival
Time Frame: 5 years
Measure: Number; unit: percentage of Patients
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
Number analyzed (Participants) | 314
percentage of Patients | 94.6

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | Accelerated Intensity Modulated Radiation Therapy (AIMRT)
All-Cause Mortality (participants affected / at risk) | 17/314
Serious Adverse Events (participants affected / at risk) | 0/314
Other Adverse Events (participants affected / at risk) | 96/314
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accelerated Intensity Modulated Radiation Therapy (AIMRT) (N=314)
Hypertension (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 2
Fatigue (General disorders) | 46
Hemolitic autoimmune anemia (Blood and lymphatic system disorders) | 1
Depression (Nervous system disorders) | 1
PAIN lower extremities (Nervous system disorders) | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
MASTITIS (Infections and infestations) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4
RASH BOTH BREASTS (Skin and subcutaneous tissue disorders) | 1
PAIN Breast Left superior aspect (Nervous system disorders) | 1
Eczema at right inframammary breast (Skin and subcutaneous tissue disorders) | 1
WEIGHT GAIN (General disorders) | 1
DERMATITIS HANDS AND FEET (Skin and subcutaneous tissue disorders) | 1 — Second Malignancy Globular ca in situ with Pagetoid spread in controlateral breast
PEDAL EDEMA (Cardiac disorders) | 1
PAIN RIGHT SHOULDER+ LEFT HIP (Nervous system disorders) | 1
RASH FUNGAL - LEFT AXILLA (Skin and subcutaneous tissue disorders) | 1
SYNCOPAL EPISODE (Cardiac disorders) | 1
Hot flashes (Endocrine disorders) | 42
DERMATITIS HANDS AND FEET (Skin and subcutaneous tissue disorders) | 1
RIGHT LEG SURGERY FOR STENT PLACEMENT (Cardiac disorders) | 1 — Cardiovascular / General Other: RIGHT LEG SURGERY FOR STENT PLACEMENT
Pain ARTHRALGIA (Nervous system disorders) | 1
ARTHRITIS LEG PAIN (Musculoskeletal and connective tissue disorders) | 1 — ARTHRITIS LEG PAIN+ CLAUDICATIO INTERMITTENS
MIGRAINE (Nervous system disorders) | 1
PAIN BACK (Nervous system disorders) | 1
CELLULITIS RIGHT ARM (Infections and infestations) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
HAIR THINNING (Skin and subcutaneous tissue disorders) | 1
MELANOMA IN SITU RIGTH LEG (Blood and lymphatic system disorders) | 1 — MELANOMA IN SITU RIGTH LEG
ADRENAL CORTICAL ADENOMA (Endocrine disorders) | 1
ACUTE APPENDICITIS (Metabolism and nutrition disorders) | 1
DEGENERATIVE SPONDILOSIS (Musculoskeletal and connective tissue disorders) | 1 — Musculoskeletal Other: DEGENERATIVE SPONDILOSIS
PAIN LEFT BREAST AT INCISION SITE sore (Nervous system disorders) | 1 — PAIN LEFT BREAST AT INCISION SITE sore
HEADACHE (Nervous system disorders) | 1 — HEADACHE
PRURITIS AT BREAST (Skin and subcutaneous tissue disorders) | 1
Pain ARTHRALGIA GENERALIZED (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1 — DIZZINESS
PAIN BACK (Nervous system disorders) | 1 — PAIN BACK
NAUSEA (Gastrointestinal disorders) | 1 — NAUSEA
PAIN AXILLA BOTH (Nervous system disorders) | 1 — PAIN AXILLA BOTH
PAIN LEFT SHOULDER (Nervous system disorders) | 1 — PAIN LEFT SHOULDER
ARTHRALGIA (Nervous system disorders) | 1 — Pain ARTHRALGIA
INCREASED LIVER ENZYMES (Hepatobiliary disorders) | 1 — INCREASED LIVER ENZYMES
FRACTURE 2ND LEFT RIB (Musculoskeletal and connective tissue disorders) | 1 — FRACTURE 2ND LEFT RIB
PAIN RIGHT THIGH (Nervous system disorders) | 1 — PAIN RIGHT THIGH
NUMBNESS (Nervous system disorders) | 1 — PINS AND NEEDLES /NUMBNESS AT SENTINEL NODES SITE
PAIN LEFT BREAST (Nervous system disorders) | 1 — PAIN LEFT BREAST ON DEEP PALPATION
Second Malignancy Invasive ductal ca (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Second Malignancy Invasive ductal ca of controlateral breast (RB)
LEFT FRACTURE ARM LEFT (Musculoskeletal and connective tissue disorders) | 1
PAIN BREAST (Nervous system disorders) | 1
PAIN BACK LOWER (Nervous system disorders) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
LYMPHEDEMA ARM LEFT (Immune system disorders) | 1
MENINGIOMA (Nervous system disorders) | 1
Secondary malignancySKIN CANCER (LEG) (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Endocrine disorders) | 1 — NIGHT SWEATS
MEMORY LOSS/UNSTEADINESS (DUE TO MENINGIOMA) (Nervous system disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
SEBORRHOIC KERATOSIS UNDER RIGHT BREAST (Skin and subcutaneous tissue disorders) | 1
PAIN BONE (Endocrine disorders) | 1 — Hot flashes
PAIN BONE (Nervous system disorders) | 1
Second Malignancy NEW PRIMARY AT LEFT BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Second Malignancy NEW PRIMARY AT LEFT BREAST
PAIN ARM LEFT (Nervous system disorders) | 1
PAIN LEFT SHOULDER (Nervous system disorders) | 1
Pain ARTHRALGIA (Nervous system disorders) | 1 — Pain ARTHRALGIA
MYALGIA (Nervous system disorders) | 1 — MYALGIA
PAIN SCAR (Nervous system disorders) | 1 — PAIN SCAR
PRURITUS (Skin and subcutaneous tissue disorders) | 1 — PRURITUS
Second Malignancy RIGHT ANKLE MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Second Malignancy RIGHT ANKLE MELANOMA
WEIGHT GAIN (General disorders) | 1 — WEIGHT GAIN
JOINT STIFFNESS, CARPAL TUNNEL SYNDROME (Musculoskeletal and connective tissue disorders) | 1 — JOINT STIFFNESS, CARPAL TUNNEL SYNDROME
PAIN Arthralgia KNEE B/L (Nervous system disorders) | 1 — PAIN Arthralgia KNEE B/L
WEIGHT LOSS (General disorders) | 1
PARESTHESIA ARM LEFT (Nervous system disorders) | 1 — PARESTHESIA ARM LEFT
Pain ARTHRALGIA - Occasional (Nervous system disorders) | 1 — Pain ARTHRALGIA - Occasional
PAIN BACK LOWER (Nervous system disorders) | 1 — PAIN BACK LOWER
PAIN RIGHT RIB AREA (Nervous system disorders) | 1 — PAIN RIGHT RIB AREA
Cardiovascular / General Other: SPLENIC HEMANGIOMA (Cardiac disorders) | 1 — Cardiovascular / General Other: SPLENIC HEMANGIOMA
HAIR THINNING (General disorders) | 1 — HAIR THINNING
PAIN RIGHT THUMB severe (Nervous system disorders) | 1 — PAIN RIGHT THUMB severe
ARTHRITIS RIGHT WRIST (Musculoskeletal and connective tissue disorders) | 1 — ARTHRITIS RIGHT WRIST

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No